CLINICAL TRIAL: NCT03803930
Title: Comparing of a 22G EUS Procore Fine Needle Biopsy Device and a 20G EUS Procore Fine Needle Biopsy Device for Solid Pancreatic Lesions: a Prospective Multi-center, Randomized, and Controlled Trial
Brief Title: Comparing of a 22G EUS Procore Fine Needle Biopsy Device and a 20G EUS Procore Fine Needle Biopsy Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: FNB20
Record Dates: First submitted 2018-12-25; First posted 2019-01-15 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Pancreas Neoplasms
Keywords: EUS-FNB; slow pull; modified wet suction technique
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 22G+SP (Other): Using 22G FNB, the first pass is SP and the pass sequence is SP-MWST-SP-MWST.
  Interventions: Device: Using 22G FNB, the first pass is SP
- Arm 22G+MWST (Other): Using 22G FNB, the first pass is MWST and the pass sequence is MWST-SP-MWST-SP.
  Interventions: Device: Using 22G FNB, the first pass is MWST
- Arm 20G+SP (Other): Using 20G FNB, the first pass is SP and the pass sequence is SP-MWST-SP-MWST.
  Interventions: Device: Using 20G FNB, the first pass is SP
- Arm 20G+MWST (Other): Using 20G FNB, the first pass is MWST and the pass sequence is MWST-SP-MWST-SP.
  Interventions: Device: Using 20G FNB, the first pass is MWST

INTERVENTIONS:
Device: Using 22G FNB, the first pass is SP — Using 22G FNB, the first pass is SP and the pass sequence is SP-MWST-SP-MWST.
  Arms: Arm 22G+SP
Device: Using 22G FNB, the first pass is MWST — Using 22G FNB, the first pass is MWST and the pass sequence is MWST-SP-MWST-SP.
  Arms: Arm 22G+MWST
Device: Using 20G FNB, the first pass is SP — Using 20G FNB, the first pass is SP and the pass sequence is SP-MWST-SP-MWST.
  Arms: Arm 20G+SP
Device: Using 20G FNB, the first pass is MWST — Using 20G FNB, the first pass is MWST and the pass sequence is MWST-SP-MWST-SP.technique-slow pull.
  Arms: Arm 20G+MWST

SUMMARY:
The purpose of this study is to compare the diagnosis accuracy of 22G EUS Procore fine needle biopsy （FNB）device and 20G EUS Procore fine needle biopsy device for solid pancreatic lesions.

DETAILED DESCRIPTION:
This is a single-blind, randomized, controlled trial. One thousand two hundred and twenty four patients with solid pancreatic lesions referred for EUS guided fine needle biopsy will be randomly assigned to 4 arms. For arm A1 which will be used with 22G EUS Procore fine needle biopsy device, the pass sequence is slow pull(SP)-modified wet suction technique(MWST)-slow pull(SP)-modified wet suction technique(MWST). For arm A2 with 22G EUS Procore fine needle biopsy device, the pass sequence is MWST-SP-MWST-SP. For arm B1 with 20G EUS Procore fine needle biopsy device, the pass sequence is SP-MWST-SP-MWST. For arm B2 with 20G EUS Procore fine needle biopsy device, the pass sequence is MWST-SP-MWST-SP. All procedures will be performed by experienced echoendoscopists, and the patients and assessors (cytologists and pathologists) will be blinded during the entire study. The primary outcome measure is the diagnosis yield. Secondary outcome measures are specimen quality.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old,<85 years old;
2. Gender: Male or Female;
3. Presence solid occupying pancreatic lesions (the diameter>1cm);
4. Must be able to receive examinations in the research center;
5. Must be able to sign the informed consent.

Exclusion Criteria:

1. Hemoglobin≤8.0 g/dl;
2. Pregnant women;
3. Coagulation disorders;
4. Took anticoagulants such as aspirin, warfarin in the latest week;
5. Acute pancreatitis in the past two weeks;
6. Cardiopulmonary dysfunction;
7. Cannot sign the informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
The diagnostic yields | up to 15 months
  The investigators' primary outcome measure is to compare the diagnostic yields of 22G FNB and 20G FNB to the solid pancreatic lesions.

SECONDARY OUTCOMES:
the tissue integrity | up to 15 months
  The investigators' secondary outcome measure is to assess the tissue size under a light microscope to compare the tissue obtained by 22G FNB and 20G FNB with Slow-pull or modified wet suction technique.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Principal Investigator — Tongji Hospital
Locations (1):
- Bin Cheng, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] DeWitt J, Jowell P, Leblanc J, McHenry L, McGreevy K, Cramer H, Volmar K, Sherman S, Gress F. EUS-guided FNA of pancreatic metastases: a multicenter experience. Gastrointest Endosc. 2005 May;61(6):689-96. doi: 10.1016/s0016-5107(05)00287-7. PMID 15855973
- [Result] Bang JY, Hebert-Magee S, Trevino J, Ramesh J, Varadarajulu S. Randomized trial comparing the 22-gauge aspiration and 22-gauge biopsy needles for EUS-guided sampling of solid pancreatic mass lesions. Gastrointest Endosc. 2012 Aug;76(2):321-7. doi: 10.1016/j.gie.2012.03.1392. Epub 2012 May 31. PMID 22658389
- [Result] Ge N, Zhang S, Jin Z, Sun S, Yang A, Wang B, Wang G, Xu G, Hao J, Zhong L, Zhong N, Li P, Zhu Q, Nian W, Li W, Zhang X, Zhou X, Yang X, Cui Y, Ding Z. Clinical use of endoscopic ultrasound-guided fine-needle aspiration: Guidelines and recommendations from Chinese Society of Digestive Endoscopy. Endosc Ultrasound. 2017 Mar-Apr;6(2):75-82. doi: 10.4103/eus.eus_20_17. No abstract available. PMID 28440232
- [Result] Gleeson FC, Kipp BR, Caudill JL, Clain JE, Clayton AC, Halling KC, Henry MR, Rajan E, Topazian MD, Wang KK, Wiersema MJ, Zhang J, Levy MJ. False positive endoscopic ultrasound fine needle aspiration cytology: incidence and risk factors. Gut. 2010 May;59(5):586-93. doi: 10.1136/gut.2009.187765. PMID 20427392
- [Result] Cheng B, Zhang Y, Chen Q, Sun B, Deng Z, Shan H, Dou L, Wang J, Li Y, Yang X, Jiang T, Xu G, Wang G. Analysis of Fine-Needle Biopsy vs Fine-Needle Aspiration in Diagnosis of Pancreatic and Abdominal Masses: A Prospective, Multicenter, Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1314-1321. doi: 10.1016/j.cgh.2017.07.010. Epub 2017 Jul 19. PMID 28733257
- [Result] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127
- [Result] Villa NA, Berzosa M, Wallace MB, Raijman I. Endoscopic ultrasound-guided fine needle aspiration: The wet suction technique. Endosc Ultrasound. 2016 Jan-Feb;5(1):17-20. doi: 10.4103/2303-9027.175877. PMID 26879162